CLINICAL TRIAL: NCT02914184
Title: Immunogenicity and Safety Study of Two Formulations of GlaxoSmithKline (GSK) Biologicals' Human Rotavirus (HRV) Vaccine (444563), in Healthy Infants Starting at Age 6-12 Weeks
Brief Title: Evaluation of Immunogenicity and Safety of Two Formulations of GSK Biologicals' Human Rotavirus (HRV) Vaccine (444563), in Healthy Infants Starting at Age 6-12 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115461; 2016-000598-19 (EudraCT Number)
Record Dates: First submitted 2016-09-16; First posted 2016-09-26 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Infections, Rotavirus; Rotavirus Vaccines
Keywords: Safety; Healthy infants; Immunogenicity; Human Rotavirus (HRV)
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Liq_A Group (Experimental): All subjects will receive two doses of PCV-free HRV liquid formulation lot A, at 6 and 12 weeks of age
  Interventions: Biological: HRV PCV-free liquid vaccine
- Liq_B Group (Experimental): All subjects will receive two doses of PCV-free HRV liquid formulation lot B, at 6 and 12 weeks of age
  Interventions: Biological: HRV PCV-free liquid vaccine
- Liq_C Group (Experimental): All subjects will receive two doses of PCV-free HRV liquid formulation lot C, at 6 and 12 weeks of age
  Interventions: Biological: HRV PCV-free liquid vaccine
- Lyo Group (Active Comparator): All subjects will receive two doses of currently licensed lyophilised HRV vaccine, at 6 and 12 weeks of age
  Interventions: Biological: Rotarix

INTERVENTIONS:
Biological: HRV PCV-free liquid vaccine — Subjects will receive two doses of PCV-free HRV vaccine at 6 and 12 weeks of age. The vaccine will be administered orally
  Arms: Liq_A Group; Liq_B Group; Liq_C Group
Biological: Rotarix — Subjects will receive two doses of currently licensed lyophilised HRV vaccine at 6 and 12 weeks of age. The vaccine will be administered orally
  Arms: Lyo Group

SUMMARY:
The purpose of this study is to evaluate the clinical consistency of three production lots of the Porcine circovirus (PCV)-free liquid formulation of oral live attenuated human rotavirus (HRV) vaccine and to evaluate the PCV-free liquid formulation of HRV vaccine as compared to the currently licensed lyophilised formulation of the HRV vaccine in terms of immunogenicity, reactogenicity and safety when administered as a two-dose vaccination in healthy infants starting at age 6-12 weeks. No new subjects will be enrolled in the extension phase of the study.

DETAILED DESCRIPTION:
* Experimental design: Phase IIIA, observer-blind, randomised (1:1:1:1), controlled, multi-centric, with four parallel groups and a staggered enrolment (Part A and Part B).
* Duration of the study: The intended duration of the study, per subject, will be approximately 7-8 months including the 6 months of extended safety follow-up period after the last dose of HRV vaccine.

  * Epoch 001: Primary starting at Visit 1 (Day 0) and ending at the safety follow-up contact (Month 7-8).
* Primary completion Date (PCD): Visit 3 (Month 2-4).
* End of Study (EoS): Last testing results released of samples collected at Visit 3 or Last Subject Last Visit (LSLV) (Follow up contact at month 7-8).
* Study Groups:

  * PCV-free HRV liquid formulation lot A (also referred to as Liq_A Group)
  * PCV-free HRV liquid formulation lot B (also referred to as Liq_B Group)
  * PCV-free HRV liquid formulation lot C (also referred to as Liq_C Group)
  * GSK Biologicals' currently licensed lyophilised HRV formulation (also referred to as Lyo Group)
* Control:active control-GSK Biologicals' currently licensed lyophilised HRV vaccine
* Vaccination schedule: Two doses of HRV vaccine to be administered according to a 0, 1-2 month schedule according to the immunisation schedule for RV vaccine.

Note that as a result of internal change in data standards terminology, the study data collected was converted to cDISC and the statistical analysis plan was amended accordingly. "Day 0" in the study design was replaced by "Day 1"; consequently, "Day n" was replaced by "Day n+1". Thus, the time frames (Day 0, Day n) of Outcome Measures described in this study record are different to that denoted in the full protocol document posted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/LAR(s) who, in the opinion of the investigator can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) (Legally acceptable representatives) of the subject prior to performing any study specific procedure.
* A male or female infant between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first study vaccination.
* Born full-term (i.e., between a gestation period of 37 weeks 0 days and 41 weeks 6 days).
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day-29 to Day 0), or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone (0.5 mg/kg/day, or equivalent). Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose of vaccine administration and ending at Visit 3, with the exception of the inactivated influenza vaccine, which is allowed at any time during the study and other licensed routine childhood vaccinations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Uncorrected congenital malformation of the gastrointestinal tract that would predispose for Intussusception (IS).
* History of IS.
* Family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Major congenital defects or serious chronic illness.
* Previous vaccination against RV.
* Previous confirmed occurrence of RVGE.
* GE within 7 days preceding the study vaccine administration.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Hypersensitivity to latex.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥38.0°C/100.4°F. The preferred location for measuring temperature in this study will be the oral cavity, the axilla and the rectum.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1612 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (19):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Cheraw, South Carolina
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Marshfield, Wisconsin
- Costa Rica (2):
  - GSK Investigational Site, San José, Provincia de San José
  - GSK Investigational Site, San José
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Germany (6):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Schönau am Königssee, Bavaria
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Bramsche
- Japan (3):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- South Korea (4):
  - GSK Investigational Site, Gangwon-do
  - GSK Investigational Site, Gyeonggido
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (7):
  - GSK Investigational Site, Málaga, Andalusia
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Taiwan (4):
  - GSK Investigational Site, Hsinchu
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20392

REFERENCES:
- [Background] Salamanca de la Cueva I, Pahud B, Huang LM, Leonardi M, Garcia-Sicilia J, Cespedes J, Abdelnour A, Tamura T, Kuroki H, Chiu NC, Virta M, Kokko S, Horn M, Panzer F, Kim JH, Jin L, Moerman L, Debacq C, Parra J, Ugarte A, Bi D; Rota-081 Study Group. Immunogenicity and safety of porcine circovirus-free human rotavirus vaccine in healthy infants: a phase III, randomized trial. J Infect Dis. 2020 May 4;225(12):2106-15. doi: 10.1093/infdis/jiaa210. Online ahead of print. PMID 32365189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 66 centers in 8 countries: 2 in Costa Rica, 10 in Finland, 6 in Germany, 7 in Japan, 6 in Republic of Korea, 9 in Spain, 6 in Taiwan and 20 in the United States (US).
Pre-assignment Details: Among 1612 subjects enrolled in the study, 1600 were vaccinated and 1545 completed the study.
Groups:
- Liq_A Group: Subjects who received two doses of PCV-free HRV liquid formulation of lot A at 6 and 12 weeks of age.
- Liq_B Group: Subjects who received two doses of PCV-free HRV liquid formulation of lot B at 6 and 12 weeks of age.
- Liq_C Group: Subjects who received two doses of PCV-free HRV liquid formulation of lot C at 6 and 12 weeks of age.
- Lyo Control Group: Subjects who received two doses of currently licensed lyophilised HRV vaccine, at 6 and 12 weeks of age.
Period: Overall Study
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
Started | 400 | 396 | 402 | 402
Completed | 386 | 383 | 385 | 391
Not Completed | 14 | 13 | 17 | 11
Not completed — Lost to Follow-up | 7 | 10 | 8 | 7
Not completed — Withdrawal by Subject | 4 | 2 | 7 | 3
Not completed — Other | 1 | 0 | 0 | 0
Not completed — Migrated/moved from the study area | 2 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group | Total
Number analyzed (Participants) | 400 | 396 | 402 | 402 | 1600
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.5 (1.5) | 8.3 (1.5) | 8.4 (1.6) | 8.5 (1.5) | 8.4 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 198 | 205 | 203 | 814
  Male | 192 | 198 | 197 | 199 | 786
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 6 | 2 | 3 | 5 | 16
  Asian | 95 | 96 | 98 | 95 | 384
  Black Or African American | 6 | 9 | 13 | 13 | 41
  Native Hawaiian Or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Other | 29 | 31 | 26 | 27 | 113
  White | 263 | 258 | 262 | 262 | 1045

OUTCOME MEASURES:

1. Primary Outcome: Anti-Rota Virus (Anti-RV) Immunoglobulin A (IgA) Antibody Concentrations in the Human Rotavirus (HRV) Liquid Formulation Groups (Liq_A, Liq_B and Liq_C)
Description: Antibody concentrations against Rota Virus (RV) were determined as Geometric Mean Antibody Concentration (GMC) and expressed as Units per milliliter (U/mL).
Time Frame: At Month 2-4 (i.e. approximately 1-month or 2-months after second dose of HRV vaccine according to the immunisation schedule for RV vaccine administration in participating countries)
Population: The analysis was performed on the Per-protocol analysis set (PPS) for immunogenicity that included all subjects who received both doses of study vaccine and for whom the liquid HRV vaccine or control vaccine was administered according to protocol and for whom immunogenicity data were available at the post-vaccination sampling time point.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group
Number analyzed (Participants) | 332 | 326 | 326
U/mL | 155.7 [125.6 to 193.1] | 147.3 [118.4 to 183.3] | 175.9 [142.8 to 216.8]
Statistical Analysis 1: Comparison: Liq_A Group vs Liq_B Group; GMC Ratio of Anti-RV IgA antibody for Liq_A and Liq_B groups was calculated using ANOVA model with vaccine groups and country as fixed effects; Test type: Other — The two-sided 95% CIs for the ratio of anti RV IgA antibody GMCs should be within the [0.5; 2] clinical limit interval; ANOVA; GMC Ratio at At Month 2-4 = 1.07, 95% CI 2-sided [0.79 to 1.44]
Statistical Analysis 2: Comparison: Liq_A Group vs Liq_C Group; GMC Ratio of Anti-RV IgA antibody for Liq_A and Liq_C groups was calculated using ANOVA model with vaccine groups and country as fixed effects; Test type: Other — The two-sided 95% CIs for the ratio of anti RV IgA antibody GMCs should be within the [0.5; 2] clinical limit interval; ANOVA; GMC Ratio at At Month 2-4 = 0.88, 95% CI 2-sided [0.65 to 1.19]
Statistical Analysis 3: Comparison: Liq_B Group vs Liq_C Group; GMC Ratio of Anti-RV IgA antibody for Liq_B and Liq_C groups was calculated using ANOVA model with vaccine groups and country as fixed effects; Test type: Other — The two-sided 95% CIs for the ratio of anti RV IgA antibody GMCs should be within the [0.5; 2] clinical limit interval; ANOVA; GMC Ratio at At Month 2-4 = 0.82, 95% CI 2-sided [0.61 to 1.11]

2. Primary Outcome: Percentage of Seroconverted Subjects With RV Antibody Concentrations Above or Equal to Cut-off Value in Porcine Circovirus (PCV) -Free Liquid HRV Vaccine (Pooled HRV Liquid Group) and Control Group
Description: Seroconversion rate (SCR) was defined as the percentage of subjects who were initially seronegative (i.e., with anti-RV IgA antibody concentration less than (<) 20 U/mL before the first dose of HRV vaccine) and developed anti-RV IgA antibody concentration greater than or equal to (≥) 20 U/mL at Month 2-4 (1-2 months after dose 2). SCR was analysed using Enzyme Linked Immunosorbent Assay (ELISA).
  For this outcome measure, the three groups (Liq_A, Liq_B & Liq_C) were pooled into a single group (Liq_Pool group) as they all received PCV free-liquid HRV vaccine, and as pre-specified in the protocol, the immunological non-inferiority of the Liq_Pool group was compared to the currently licensed lyophilized HRV vaccine (Lyo_Control group) in terms of seroconversion rates of 1-2 months after Dose 2.
Time Frame: as for outcome 1
Population: The analysis was performed on the PPS for immunogenicity that included all subjects who received both doses of study vaccine and for whom the liquid HRV vaccine or control vaccine was administered according to protocol and for whom immunogenicity data were available at the post-vaccination sampling time point.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Liq_Pool Group: Subjects who received two doses of PCV-free HRV liquid formulation of pooled lot A, B and C at 6 and 12 weeks of age.
Arm/Group | Liq_Pool Group | Lyo Control Group
Number analyzed (Participants) | 984 | 329
Percentage of subjects | 79.3 [76.6 to 81.8] | 81.8 [77.2 to 85.8]
Statistical Analysis 1: Comparison: Liq_Pool Group vs Lyo Control Group; Non-inferiority of Liq_Pool group compared to Lyo Control group in terms of difference in % of subjects with anti-RV IgA titer ≥ specified cut off with its 2-sided 95% CI in initially seronegative subjects; Test type: Non-Inferiority — Lower limit (LL) of the two-sided asymptotic standardized 95% CI for the difference in SCR for antibodies to rota virus at month 2-4 between the Liq_Pool group and Lyo Control group should be ≥ -10%; SCR difference at Month 2-4 = -2.49, 95% CI 2-sided [-7.15 to 2.63]

3. Primary Outcome: Percentage of Seroconverted Subjects With RV Antibody Concentrations Above or Equal to 20 U/mL in Porcine Circovirus (PCV)-Free Liquid HRV Vaccine (Individual HRV Liquid Groups) and Lyophilised Control Group
Description: Seroconversion rate (SCR) was defined as the percentage of subjects who were initially seronegative (i.e., with anti-RV IgA antibody concentration less than (<) 20 U/mL before the first dose of HRV vaccine) and developed anti-RV IgA antibody concentration greater than or equal to (≥) 20 U/mL at Month 2-4 (1-2 months after dose 2). SCR was analysed using Enzyme Linked Immunosorbent Assay (ELISA).
  The analysis was assessed to demonstrate the immunogenicity of PCV-free liquid HRV vaccine as compared to the currently licensed lyophilised HRV vaccine (individual HRV liquid groups) in terms of seroconversion rates 1-2 months after Dose 2.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
Number analyzed (Participants) | 332 | 326 | 326 | 329
Percentage of subjects | 77.7 [72.8 to 82.1] | 77.6 [72.7 to 82.0] | 82.5 [77.9 to 86.5] | 81.8 [77.2 to 85.8]

4. Primary Outcome: Anti-RV IgA Antibody Concentrations in the PCV-free Liquid HRV Vaccine (Pooled HRV Liquid Group) and Lyophilised Control Group
Description: Antibody concentrations against RV were determined as GMCs and expressed as U/mL.
  For this outcome measure, the three groups (Liq_A, Liq_B & Liq_C) were pooled into a single group (Liq_Pool group) as they all received PCV free-liquid HRV vaccine, and as pre-specified in the protocol, the immunological non-inferiority of the Liq_Pool group was compared to the currently licensed lyophilized HRV vaccine (Lyo_Control group) in terms of antibody concentrations at 1-2 months after Dose 2.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Liq_Pool Group | Lyo Control Group
Number analyzed (Participants) | 984 | 329
U/mL | 159.2 [140.7 to 180.1] | 153.8 [125.1 to 189.0]
Statistical Analysis 1: Comparison: Liq_Pool Group vs Lyo Control Group; Non-inferiority of Liq_Pool Group as compared to Lyo Control group in terms of the GMC ratio calculated using ANOVA model with vaccine groups and country as fixed effects; Test type: Non-Inferiority — LL of the two-sided 95% CI for the ratio of anti-RV IgA antibody GMCs between the Liq_Pool Group and Control group should be ≥ 0.67; ANOVA; GMC Ratio at At Month 2-4 = 1.04, 95% CI 2-sided [0.82 to 1.33]

5. Primary Outcome: Anti-RV IgA Antibody Concentrations in the PCV-free Liquid HRV Vaccine (Individual HRV Liquid Groups) and Lyophilised Control Group
Description: Antibody concentrations against RV were determined as GMCs and expressed as U/mL. The analysis was assessed to demonstrate the immunogenicity of the PCV-free liquid HRV vaccine (individual HRV liquid groups) to that of the currently licensed lyophilised HRV vaccine in terms of serum anti-RV IgA antibody concentrations 1-2 months after Dose 2.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
Number analyzed (Participants) | 332 | 326 | 326 | 329
U/mL | 155.7 [125.6 to 193.1] | 147.3 [118.4 to 183.3] | 175.9 [142.8 to 216.8] | 153.8 [125.1 to 189.0]

6. Secondary Outcome: Percentage of Subjects With Anti-RV IgA Concentrations (Pooled HRV Liquid Group)
Description: Antibody concentrations ≥90 U/mL were determined and expressed as GMCs, assessed for the pooled HRV liquid groups and Control Group. The GMC calculations were performed by taking the anti-log of the mean of the log concentration transformations.
  For this outcome measure, the three groups (Liq_A, Liq_B & Liq_C) were pooled into a single group (Liq_Pool group) as they all received PCV free-liquid HRV vaccine, and as pre-specified in the protocol, the immunogenicity of the Liq_Pool group was compared to the currently licensed lyophilized HRV vaccine (Lyo_Control group) in terms of percentage of subjects with anti-RV IgA antibody concentrations ≥ 90 U/mL, 1-2 months after Dose 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Liq_Pool Group | Lyo Control Group
Number analyzed (Participants) | 984 | 329
Percentage of subjects | 63.0 [59.9 to 66.0] | 62.3 [56.8 to 67.6]

7. Secondary Outcome: Percentage of Subjects With Anti-RV IgA Concentrations (Individual HRV Liquid Groups)
Description: Antibody concentrations ≥90 U/mL were determined and expressed as GMCs, assessed for the individual HRV liquid groups and Control Group. The GMC calculations were performed by taking the anti-log of the mean of the log concentration transformations. The analysis was performed to assess the immunogenicity of the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and the currently licensed lyophilised HRV vaccine, in terms of percentage of subjects with anti-RV IgA antibody concentrations ≥ 90 U/mL 1-2 months after Dose 2.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
Number analyzed (Participants) | 322 | 326 | 326 | 329
Percentage of subjects | 62.7 [57.2 to 67.9] | 61.0 [55.5 to 66.4] | 65.3 [59.9 to 70.5] | 62.3 [56.8 to 67.6]

8. Secondary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs).
Description: Assessed solicited general AEs were cough/runny nose, diarrhea, fever (defined as temperature ≥ 38.0°C), irritability/fussiness, loss of appetite and vomiting. Any solicited general AE is defined as any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination.
Time Frame: During the 8 days (Day 1 to Day 8) follow-up period after each dose of HRV vaccine
Population: Analysis was performed on the Exposed Set (ES). The ES included all subjects with at least one study vaccine administration documented. A safety analysis based on the ES included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
Number analyzed (Participants) | 400 | 396 | 402 | 402
Participants
  Any - Cough / Runny Nose - Dose 1 | 93 | 91 | 94 | 102
  Any - Cough / Runny Nose - Dose 2: number analyzed (Participants) | 393 | 396 | 392 | 394
  Any - Cough / Runny Nose - Dose 2 | 114 | 100 | 94 | 109
  Any - Diarrhea - Dose 1 | 14 | 13 | 8 | 10
  Any - Diarrhea - Dose 2: number analyzed (Participants) | 393 | 396 | 392 | 394
  Any - Diarrhea - Dose 2 | 7 | 12 | 8 | 11
  Any - Fever (≥ 38.0°C) - Dose 1 | 24 | 22 | 20 | 23
  Any - Fever (≥ 38.0°C) - Dose 2: number analyzed (Participants) | 393 | 396 | 392 | 394
  Any - Fever (≥ 38.0°C) - Dose 2 | 36 | 36 | 34 | 32
  Any - Irritability / Fussiness - Dose 1 | 226 | 214 | 209 | 216
  Any - Irritability / Fussiness - Dose 2: number analyzed (Participants) | 393 | 396 | 392 | 394
  Any - Irritability / Fussiness - Dose 2 | 191 | 189 | 194 | 194
  Any - Loss of appetite - Dose 1 | 97 | 93 | 99 | 96
  Any - Loss of appetite - Dose 2: number analyzed (Participants) | 393 | 396 | 392 | 394
  Any - Loss of appetite - Dose 2 | 92 | 84 | 78 | 94
  Any - Vomiting - Dose 1 | 39 | 51 | 38 | 42
  Any - Vomiting - Dose 2: number analyzed (Participants) | 393 | 396 | 392 | 394
  Any - Vomiting - Dose 2 | 25 | 28 | 31 | 34

9. Secondary Outcome: Number of Subjects With Any Unsolicited AEs.
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any is defined as the occurrence of any unsolicited AE irrespective of its intensity grade and relationship to vaccination.
Time Frame: During the 31 day (Day 1 to Day 31) follow-up period after HRV vaccination across doses
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
Number analyzed (Participants) | 400 | 396 | 402 | 402
Participants | 183 | 189 | 200 | 184

10. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include any untoward medical occurrence that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity.
Time Frame: During the entire study period (Day 1 to Month 7-8)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
Number analyzed (Participants) | 400 | 396 | 402 | 402
Participants | 21 | 18 | 21 | 18

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 8 days (Day 1 to Day 8) follow-up period after each vaccination. Unsolicited AEs: During the 31 days (Day 1 to Day 31) follow-up period after vaccination. SAEs: Throughout the study period (Day 1 to Month 7-8).
Arm/Group | Liq_A Group | Liq_B Group | Liq_C Group | Lyo Control Group
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/396 | 0/402 | 0/402
Serious Adverse Events (participants affected / at risk) | 21/400 | 18/396 | 21/402 | 18/402
Other Adverse Events (participants affected / at risk) | 333/400 | 242/396 | 338/402 | 338/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liq_A Group (N=400) | Liq_B Group (N=396) | Liq_C Group (N=402) | Lyo Control Group (N=402)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 4 (4) | 3 (3) | 3 (4) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Encephalitis enteroviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infantile spasms (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 6 (6) | 6 (6) | 3 (3) | 2 (2)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liq_A Group (N=400) | Liq_B Group (N=396) | Liq_C Group (N=402) | Lyo Control Group (N=402)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brachycephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gray matter heterotopia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plagiocephaly (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 3 (3) | 5 (5) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (8) | 10 (10) | 4 (5) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 38 (57) | 25 (25) | 31 (45) | 44 (59)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (7) | 3 (3) | 4 (5) | 8 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 9 (9) | 4 (4) | 11 (11)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Infantile colic (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (7) | 6 (6) | 3 (3) | 2 (2)
Crying (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 10 (10) | 8 (8) | 13 (13) | 6 (6)
Vaccination site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 3 (3) | 1 (1) | 1 (2) | 4 (4)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 10 (10) | 10 (10) | 7 (7) | 9 (9)
Bronchitis (Infections and infestations) | 5 (5) | 4 (4) | 6 (6) | 4 (4)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 7 (7) | 5 (5) | 11 (11) | 11 (12)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (9) | 6 (6) | 3 (5) | 3 (5)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 6 (6)
Laryngitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 24 (25) | 25 (25) | 36 (40) | 29 (37)
Oral candidiasis (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 8 (8)
Oral fungal infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 5 (5) | 4 (4) | 2 (2)
Otitis media acute (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 5 (5)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (3) | 8 (8) | 4 (4) | 8 (9)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 3 (5) | 7 (7) | 6 (6) | 6 (6)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subglottic laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 31 (33) | 34 (34) | 31 (36) | 30 (32)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 3 (4) | 6 (6)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 145 (192) | 0 (0) | 139 (177) | 141 (191)
Feeding disorder (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 276 (426) | 5 (5) | 264 (408) | 261 (419)
Merycism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Selective eating disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crystalluria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile adhesion (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 165 (213) | 6 (6) | 152 (198) | 163 (214)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 2 (2) | 5 (5)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 6 (6) | 2 (3)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 3 (3) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 9 (9) | 4 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 8 (10) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 9 (10) | 3 (3) | 8 (8) | 7 (8)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 4 (4)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT02914184/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT02914184/SAP_001.pdf